CLINICAL TRIAL: NCT03068819
Title: Cytokine Induced Memory-like NK Cell Adoptive Therapy for Relapsed AML After Allogeneic Hematopoietic Cell Transplant in Children and Adults
Brief Title: Cytokine Induced Memory-like NK Cell Adoptive Therapy for Relapsed AML After Allogeneic Hematopoietic Cell Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Wugen, Inc. (Industry); Children's Discovery Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202206197; P50CA171963 (NIH)
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CIML NK cell after T cell DLT (Pilot Pediatric/Young Adult Cohort) (Experimental): * The recipient will receive standard of care salvage chemotherapy consisting of fludarabine (or cladribine if shortage), cytarabine, and G-CSF (FLAG) to be started 2 to 4 weeks prior to the CIML NK cell infusion. 5-day decitabine is an acceptable alternative for FLAG, and another standard of care salvage chemotherapy regimen, if clinically appropriate and approved by the study PI, may be used.
  * The donor will undergo non-mobilized leukapheresis on Day -2 or -1. Standard of care DLI (1 x 10^6 CD3+ cells/kg) will be given fresh on day -1.
  * A second cycle of therapy may be administered > 30 days after the administration of the first course of protocol therapy to maintain response or to treat persistent/relapsed AML, if a patient continues to meet the inclusion/exclusion criteria. Chemotherapy may be omitted before a second infusion of DLI and CIML NK cells. In the setting of GVHD following the first cycle of therapy, the T cell DLI may be omitted, and ML NK cells administered.
  Interventions: Drug: CIML NK Cell Infusion; Procedure: CD3+ T Cell Product Infusion
- CIML NK cell after T cell DLT (Phase 2 Adult Cohort) (Experimental): * The recipient will receive lymphodepleting chemotherapy with fludarabine (or cladribine if shortage) and cyclophosphamide beginning on day -7.
  * The donor will undergo non-mobilized leukapheresis on Day -2 or -1. T cell dose per standard of care institutional practices and physician discretion will be given frozen for administration on day 30.
  * A second cycle of therapy may be administered > 30 days after the administration of the first course of protocol therapy to maintain response or to treat persistent/relapsed AML, if a patient continues to meet the inclusion/exclusion criteria. Chemotherapy may be omitted before a second infusion of DLI and CIML NK cells. In the setting of GVHD following the first cycle of therapy, the T cell DLI may be omitted, and ML NK cells administered. The date of the second NK cell infusion will be considered a second Day 0.
  Interventions: Drug: CIML NK Cell Infusion; Procedure: CD3+ T Cell Product Infusion

INTERVENTIONS:
Drug: CIML NK Cell Infusion — -Day 0
Procedure: CD3+ T Cell Product Infusion — -Day -1

SUMMARY:
Donor Lymphocyte Infusion (DLI) following salvage chemotherapy is the one of the most widely used treatment approaches in patients who relapse after allogeneic hematopoietic cell transplant (allo-HCT). However, the complete remission (CR) rates and long term survival remain very poor in these patients and, therefore, there is an unmet need to develop more effective treatment approaches in patients who relapse after allo-HCT.

Based on the initial promising results with our ongoing cytokine-induced memory-like (CIML) natural killer (NK) cell trial, the investigators hypothesize that combining the CIML NK cells with DLI approach will significantly enhance the graft versus leukemia and therefore potentially provide potentially curative therapy for these patients with otherwise extremely poor prognosis. Combining CIML NK cells with the DLI platform will also potentially allow these adoptively transferred cells to persist for longer duration as they should not be rejected by donor T cells as the CIML NK cells are derived from the same donor. The use of CIML NK cells is unlikely to lead to excessive graft versus host disease (GVHD) as previous studies have not been associated with excessive GVHD rates.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Relapsed AML after HLA-matched related or unrelated allogeneic hematopoietic cell transplant
* For pilot pediatric/young adult patient cohort ≥1 and <18 years of age
* For phase 2 adult patient cohort ≥18 years of age
* Available original donor (same donor as used for the initial stem cell transplant) that is willing and eligible for non-mobilized collection
* Patients with known central nervous system (CNS) involvement with AML are eligible provided that they have been treated and cerebrospinal fluid (CSF) is clear for at least 2 weeks prior to enrollment into the study. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the study treatment.
* Karnofsky performance status > 60 %
* Adequate organ function as defined below:

  * Total bilirubin < 2 mg/dL
  * AST(SGOT)/ALT(SGPT) < 3.0 x IULN
  * Creatinine within normal institutional limits OR creatinine clearance > 60 mL/min/1.73 m2 by Cockcroft-Gault Formula
  * Oxygen saturation ≥90% on room air
* Not currently requiring systemic corticosteroid therapy (10 mg or less of prednisone or equivalent doses of other systemic steroids are allowed) or any other immune suppressive medications
* Women of childbearing potential must have a negative pregnancy test within 28 days prior to study registration. Female and male patients (along with their female partners) must agree to use two forms of acceptable contraception, including one barrier method, during participation in the study including throughout the initial evaluation period (100 days after CIML NK cell infusion).
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Recipient Exclusion Criteria:

* Acute or chronic GvHD with ongoing active systemic treatment.
* Circulating blast count >10,000/uL by morphology or flow cytometry (cyto-reductive therapies, including salvage chemotherapy, is encouraged prior to study enrollment)
* Uncontrolled bacterial or viral infections, or known HIV, Hepatitis B, or Hepatitis C infection.
* Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or EKG suggestive of acute ischemia or active conduction system abnormalities.
* New or progressive pulmonary infiltrates concerning for new or uncontrolled infectious process.
* Known hypersensitivity to one or more of the study agents
* Received any investigational drugs within the 14 days prior to CIML NK cell infusion date
* Pregnant and/or breastfeeding

Donor Inclusion Criteria:

* At least 18 years of age
* Same donor as used for the allo-HCT
* In general good health, and medically able to tolerate leukapheresis
* Ability to understand and willingness to sign an IRB approved written informed consent document

Donor Exclusion Criteria:

* Active hepatitis, positive for HTLV, or HIV on donor viral screen
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of regimen defined as the number of participants who are successfully infused with T cell DLT and CIML NK cells (Pilot Pediatric/Young Adult Cohort) | Completion of all patients through Day 0 (estimated to be 102 months)
  -Will be considered successful if doses above the minimum can be delivered in at least 18 of 24 patients. Target and minimum CIML doses are maximum capped at 20x10^6/kg with a minimum dose of 0.5x10^6 kg.
Safety of administering CIML NK cells plus T cell DLT as measured by unexpected early mortality (Pilot Pediatric/Young Adult Cohort) | Up to Day 100
Safety of administering CIML NK cells plus T cell DLT as measured by excess acute or chronic GVHD (Pilot Pediatric/Young Adult Cohort) | Up to 12 months
Safety of administering CIML NK cells plus T cell DLT as measured by prolonged neutropenia (Pilot Pediatric/Young Adult Cohort) | 8 weeks post CIML NK infusion
Safety of administering CIML NK cells plus T cell DLT as measured by unexpected early mortality (Phase 2 Adult Cohort) | Up to Day 100
  -Patients will be continually assessed for unexpected early mortality (as assessed at Day +30 and Day +100 after CIML NK cell infusion), associated with the study treatment.
Safety of administering CIML NK cells plus T cell DLT as measured by unacceptable GVHD (Phase 2 Adult Cohort) | Up to 12 months
Safety of administering CIML NK cells plus T cell DLT as measured by prolonged neutropenia (Phase 2 Adult Cohort) | 8 weeks post CIML NK infusion
Rate of leukemia-free survival (LFS) (Phase 2 Adult Cohort) | 6 months
  -LFS is defined as the time from achievement of CR/CRi to the time of relapse, death in remission, or last follow-up.

SECONDARY OUTCOMES:
Complete remission rate (CR/CRi) (Pilot Pediatric/Young Adult Cohort) | Day 30
  * Complete remission (CR):Morphologically leukemia free state (i.e. bone marrow with <5% blasts by morphologic criteria and no blasts with Auer rods, no evidence of extramedullary leukemia) and absolute neutrophil count ≥1000 /μL and platelets ≥100,000 /μL. Patient must be independent of transfusions
  * Complete remission with incomplete blood count recover (CRi): All of the above criteria for CR must be met, except that absolute neutrophils <1000 /μL or platelets <100,000 /μL in the blood.
Rate of leukemia-free survival (LFS) (Pilot Pediatric/Young Adult Cohort) | 100 days post CIML NK cell infusion
  -LFS is defined as the time from achievement of CR/CRi to the time of relapse, death in remission, or last follow-up.
Overall survival (OS) (Pilot Pediatric/Young Adult Cohort) | 100 days post CIML NK cell infusion
  -OS is defined as the time from the date of Day 0 until death from any cause.
Rate of leukemia-free survival (LFS) (Pilot Pediatric/Young Adult Cohort) | 1 year post CIML NK cell infusion
  -LFS is defined as the time from achievement of CR/CRi to the time of relapse, death in remission, or last follow-up.
Overall survival (OS) (Pilot Pediatric/Young Adult Cohort) | 1 year post CIML NK cell infusion
  -OS is defined as the time from the date of Day 0 until death from any cause.
Incidence and severity of acute GVHD rates (Pilot Pediatric/Young Adult Cohort) | Day 14 through 6 months
  -Incidence and severity of acute GVHD will be assessed based on the Minnesota grading scale. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).
Incidence and severity of acute GVHD rates (Pilot Pediatric/Young Adult Cohort) | Day 14 through 6 months
  -Incidence and severity of acute GVHD will be assessed based on the CIBMTR grading scale. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).
Incidence and severity of chronic GVHD rates (Pilot Pediatric/Young Adult Cohort) | Day 100 through 12 months
  -Incidence and severity of chronic GVHD will be assessed based on the NIH consensus criteria and global severity scoring system. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).
Complete remission rate (CR/CRi) (Phase 2 Adult Cohort) | Day 30
  * Complete remission (CR):Morphologically leukemia free state (i.e. bone marrow with <5% blasts by morphologic criteria and no blasts with Auer rods, no evidence of extramedullary leukemia) and absolute neutrophil count ≥1000 /μL and platelets ≥100,000 /μL. Patient must be independent of transfusions
  * Complete remission with incomplete blood count recover (CRi): All of the above criteria for CR must be met, except that absolute neutrophils <1000 /μL or platelets <100,000 /μL in the blood.
Rate of leukemia-free survival (LFS) (Phase 2 Adult Cohort) | 100 days post CIML NK cell infusion
  -LFS is defined as the time from achievement of CR/CRi to the time of relapse, death in remission, or last follow-up.
Overall survival (OS) (Phase 2 Adult Cohort) | 100 days post CIML NK cell infusion
  -OS is defined as the time from the date of Day 0 until death from any cause.
Rate of leukemia-free survival (LFS) (Phase 2 Adult Cohort) | 1 year post CIML NK cell infusion
  -LFS is defined as the time from achievement of CR/CRi to the time of relapse, death in remission, or last follow-up.
Overall survival (OS) (Phase 2 Adult Cohort) | 1 year post CIML NK cell infusion
  -OS is defined as the time from the date of Day 0 until death from any cause.
Incidence and severity of acute GVHD rates (Phase 2 Adult Cohort) | Day 14 through 6 months
  -Incidence and severity of acute GVHD will be assessed based on the CIBMTR grading scale. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).
Incidence and severity of chronic GVHD rates (Phase 2 Adult Cohort) | Day 100 through 12 months
  -Incidence and severity of chronic GVHD will be assessed based on the NIH consensus criteria and global severity scoring system. Attempts should be made to confirm the diagnosis pathologically by biopsy of target organ(s).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cashen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bednarski JJ, Zimmerman C, Berrien-Elliott MM, Foltz JA, Becker-Hapak M, Neal CC, Foster M, Schappe T, McClain E, Pence PP, Desai S, Kersting-Schadek S, Wong P, Russler-Germain DA, Fisk B, Lie WR, Eisele J, Hyde S, Bhatt ST, Griffith OL, Griffith M, Petti AA, Cashen AF, Fehniger TA. Donor memory-like NK cells persist and induce remissions in pediatric patients with relapsed AML after transplant. Blood. 2022 Mar 17;139(11):1670-1683. doi: 10.1182/blood.2021013972. PMID 34871371
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu